CLINICAL TRIAL: NCT01113749
Title: Improving Decision Making About Feeding Options for Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 05-3105; 5R01NR009826 (NIH)
Record Dates: First submitted 2010-04-15; First posted 2010-04-30 (Estimated); Results first posted 2012-08-10 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2012-04

CONDITIONS: Dementia
Keywords: Dementia; Nutrition; Feeding
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision support (Experimental): Structured decision aid with prompting to share information in discussion with primary treating health care providers.
  Interventions: Other: Feeding Options in Dementia Decision Aid
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Feeding Options in Dementia Decision Aid — Structured decision aid on feeding options in dementia care with prompting to share information in discussion with primary treating health care provider.
  Arms: Decision support

SUMMARY:
This study is a randomized trial to test whether a decision aid can help to improve the quality of decision making about feeding options in care of patients with dementia.

DETAILED DESCRIPTION:
This research study is a cluster randomized controlled trial of a decision aid to improve decision-making about feeding options for patients with advanced dementia. Surrogate decision-makers in the nursing homes randomized to the intervention will review the decision aid and be prompted to discuss it with the primary health care provider, while those in the control sites receive usual care. We measure the immediate, 1 and 3 month effects of the decision aid on the quality of surrogate decision-making for nursing home residents with advanced dementia.

ELIGIBILITY:
Inclusion Criteria:

* dementia diagnosis
* advanced cognitive impairment
* feeding problem
* age >= 65
* surrogate decision maker

Exclusion Criteria:

* feeding tube decision made
* hospice
* BMI > 26
* major psychosis or developmental delay

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Hanson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Hanson LC, Ersek M, Lin FC, Carey TS. Outcomes of feeding problems in advanced dementia in a nursing home population. J Am Geriatr Soc. 2013 Oct;61(10):1692-7. doi: 10.1111/jgs.12448. Epub 2013 Sep 19. PMID 24083403
- [Derived] Hanson LC, Carey TS, Caprio AJ, Lee TJ, Ersek M, Garrett J, Jackman A, Gilliam R, Wessell K, Mitchell SL. Improving decision-making for feeding options in advanced dementia: a randomized, controlled trial. J Am Geriatr Soc. 2011 Nov;59(11):2009-16. doi: 10.1111/j.1532-5415.2011.03629.x. Epub 2011 Sep 15. PMID 22091750
- [Derived] Hanson LC, Gilliam R, Lee TJ. Successful clinical trial research in nursing homes: the Improving Decision-Making Study. Clin Trials. 2010 Dec;7(6):735-43. doi: 10.1177/1740774510380241. Epub 2010 Aug 20. PMID 20729251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 425 eligible dementia resident-surrogate dyads identified ; 118 surrogates refused, 41 unable to contact, and 10 unable to participate due to concurrent illness.
Pre-assignment Details: No enrolled participants were excluded before assignment
Period: Overall Study
Arm/Group | Decision Support | Control
Started | 127 | 129
Completed | 126 | 127
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Support | Control | Total
Number analyzed (Participants) | 127 | 129 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 127 | 129 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.2 (2.1) | 85.3 (2.3) | 85.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 98 | 195
  Male | 30 | 31 | 61
Region of Enrollment [Number; unit: participants]
  United States | 127 | 129 | 256

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict Scale
Description: Decisional Conflict Scale measures conflict in decisions Total scale range 1-5 with lower scores indicating less conflict.
Time Frame: 3 months
Population: intention to treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Decision Support Intervention: Decision aid
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 127 | 129
units on a scale | 1.65 (NA) [1.53 to 1.73] | 1.97 (NA) [1.86 to 2.14]

2. Secondary Outcome: Percent With Treatment Decisions
Description: Treatment decisions are expressed as percentage of subjects with discussions of new tube feeding, new orders to forego tube feeding, and new choices for assisted feeding.
Time Frame: 3 months
Measure: Number; unit: percentage of subjects
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 127 | 129
percentage of subjects | 46 [NA to NA] | 33 [NA to NA]

3. Post Hoc Outcome: Percentage of Subjects With Weight Loss
Description: Percentage of subjects with weight loss at 9 months
Time Frame: 9 months
Population: intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Decision Support Intervention | Control
Number analyzed (Participants) | 127 | 129
percentage of participants | 6 | 16

ADVERSE EVENTS:
Arm/Group | Decisions Support Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/129
Other Adverse Events (participants affected / at risk) | 0/127 | 0/129

LIMITATIONS AND CAVEATS:
Cluster randomization required, preventing double-blinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No